CLINICAL TRIAL: NCT04463186
Title: Time-based Effects of Different Duration Stretching on Calf Muscle Strength
Brief Title: Time Based Effects of Different Duration Stretching on Calf Muscle Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Masood Khan, Principal investigator, King Saud University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RRC-2019-05
Record Dates: First submitted 2020-07-05; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Muscle Strength
Keywords: Muscle strength; muscle stretching exercises; Calf Muscle
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Subjects participated in three experimental trials: Static stretching for 2 minutes (SS2), static stretching for 4 minutes (SS4), and static stretching for 8 minutes (SS8). Strength was measured before (pre), immediately after (post), and at 10- and 20- minutes post stretching.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): subjects participated in three experimental trials: Static stretching for 2 minutes (SS2), static stretching for 4 minutes (SS4), and static stretching for 8 minutes (SS8). Strength was measured before (pre), immediately after (post), and at 10- and 20- minutes post stretching.
  Interventions: Other: Muscle Static Stretching

INTERVENTIONS:
Other: Muscle Static Stretching — Static stretching for 2 minutes (SS2), static stretching for 4 minutes (SS4), and static stretching for 8 minutes (SS8). Each static stretching (SS) trial involved varied repetitions of 30-seconds self-stretches and 20-seconds relax periods.

SUMMARY:
Stretching is reported to decrease muscle strength and thus suggested to be avoided prior to athletic events but with conflicting reports. This time course study aimed to assess acute effects of static stretching of different durations on isometric maximum voluntary contraction force of calf muscle.

DETAILED DESCRIPTION:
Stretching is reported to decrease muscle strength and thus suggested to be avoided prior to athletic events but with conflicting reports. This time course study aimed to assess acute effects of static stretching of different durations on isometric maximum voluntary contraction force of calf muscle. Pretest posttest experimental design was used. 14 subjects participated in three experimental trials: Static stretching for 2 minutes (SS2), static stretching for 4 minutes (SS4), and static stretching for 8 minutes (SS8). Strength was measured before (pre), immediately after (post), and at 10- and 20- minutes post stretching. Each static stretching (SS) trial involved varied repetitions of 30-seconds self-stretches and 20-seconds relax periods.

ELIGIBILITY:
Inclusion Criteria:

* Subjects performed active foot dorsiflexion in long sitting position with back supported against wall and those having not more than 20-degree range of motion were selected
* Used to engage in 1 to 5 hours of physical activity per week

Exclusion Criteria:

* Subjects having any current injury or limits in range of motion specific to lower limb joints
* Current neuromuscular disease
* Competitive athletes were excluded from the study

Ages: 24 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Change in Isometric Maximum Voluntary Contraction Force | MVCF at baseline and 0, 10, 20-min post stretching
  Isometric Maximum Voluntary Contraction Force was measured using strain Gauge.

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided